CLINICAL TRIAL: NCT02405221
Title: A Pilot Clinical Trial Assessing the Safety and Feasibility of Intramuscular Administration of the TA-CIN Vaccine as Adjuvant Therapy for Patients With History of HPV16 Associated Cervical Cancer
Brief Title: Safety and Feasibility of TA-CIN Vaccine in HPV16 Associated Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); PapiVax Biotech, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1553; IRB00054202 (Other: JHMIRB); P50CA098252 (NIH)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: HPV16 Associated Cervical Cancer
Keywords: HPV; HPV16; Cervical Cancer; TA-CIN; Vaccine; Adjuvant; Nickles FaderPI
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TA-CIN administration via thigh (Experimental): Each dose of TA-CIN vaccine is fixed, 100µg. Patients will receive 3 doses of the TA-CIN 4 weeks apart (Weeks 1, 5, and 9), administered in the thigh. Patients will be followed for 2 years after the 1st dose is given.
  Interventions: Biological: TA-CIN (thigh)
- TA-CIN administration via arm (Experimental): Each dose of TA-CIN vaccine is fixed, 100µg. Patients will receive 3 doses of the TA-CIN 4 weeks apart (Weeks 1, 5, and 9), administered in the arm. Patients will be followed for 2 years after the 1st dose is given.
  Interventions: Biological: TA-CIN (arm)

INTERVENTIONS:
Biological: TA-CIN (arm) — TA-CIN vaccine 100µg IM in the arm at Week 1, 5, and 9.
  Other Names: Tissue Antigen - Cervical Intraepithelial Neoplasia
  Arms: TA-CIN administration via arm
Biological: TA-CIN (thigh) — TA-CIN vaccine 100µg IM in the arm at Week 1, 5, and 9.
  Other Names: Tissue Antigen - Cervical Intraepithelial Neoplasia
  Arms: TA-CIN administration via thigh

SUMMARY:
This study will be looking at what dose of the TA-CIN vaccine is safe and effective in patients with a history of HPV16-associated cervical cancer.

DETAILED DESCRIPTION:
This is a randomized, multi-center, open label pilot study. The primary goal of this study is to determine the safety of TA-CIN vaccine as adjuvant therapy, and to assess evidence of induction of HPV antigen-specific immunologic response when administered at different locations (arm or thigh). In this pilot study, a single dose level (100µg) assessment of the safety and tolerability of administering TA-CIN vaccine three times to either the arm versus the thigh of patients who have previously been treated for HPV16-related cervical cancer in the past year and are documented to have no evidence of disease recurrence based on standard-of-care imaging and/or clinical assessment upon eligibility.

A total of 14 patients will be enrolled to assess the safety of TA-CIN vaccine via different injection sites as adjuvant therapy. Safety assessments will continue for a period for 1 month after the last vaccination. Few or no serious adverse events (SAEs) are expected from this regimen and routes of administration. The motivation for the design is to confirm that the dose and site of injection implemented here has minimal or no systemic toxicity, as well as determining the preferred injection site that can elicit more potent immune response.

The study will consist of the following parts:

* Screening evaluation
* Dosing period and response assessments
* Follow-up visits after last dose

Screening Evaluation:

The screening visit will be performed within 60 days of the first study drug administration visit. The study team will check the results of these screening tests to see if patient qualifies to participate.

Dosing Period:

Those who meet the study requirements during the screening period will then begin the dosing phase of this study. TA-CIN will be given as a single intramuscular injection every 4 weeks for a maximum of 3 times. The location of the injection (arm or thigh) will depend on randomization. Patients will be assessed for safety and response to treatment during this period.

Follow-Up Period:

Four follow-up evaluations will be performed during a clinic visit after the last dose of the vaccine. These will take place at the following time points: (1) 1-3 weeks after the last dose of the study drug, (2) about 6 months after the last dose of the study drug, (3) about 12 months after the last dose of the study drug, and (4) about 24 months after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HPV16 related stage IB1-IV cervical cancer who completed definitive treatment within 12 months
2. Patients with no evidence of disease recurrence within 8 weeks of enrollment
3. Documented to have HPV16 nucleic acid within the cervical tumor specimen as determined by in situ hybridization
4. Fresh-frozen or paraffin-embedded material must be available for in situ hybridization testing for HPV16 nucleic acid for central confirmation
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
6. Adequate organ function as defined by study-specified laboratory tests
7. Ability to understand and willingness to sign a written informed consent document
8. Willing and able to comply with study schedule and other protocol requirements

Exclusion Criteria:

1. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
2. Patients with a diagnosis of immunosuppression or prolonged, active use of immunosuppressive agents such as systemic steroids
3. Prior HPV vaccination
4. Had surgery, chemotherapy, or radiation therapy within 28 days prior to receiving study drug
5. Another investigational product within 28 days prior to receiving study drug
6. Active or chronic HIV, HBV, or HCV infection
7. Pregnant or lactating
8. Patients who have an active autoimmune disease
9. Patients with a recognized immunodeficiency disease or are being chronically treated with immunosuppressive drugs
10. Women of childbearing potential
11. Patients with non-healed wounds
12. A history of current or recent concurrent malignancy (≤5 years) except basal cell cancer.
13. Inability to understand or unwillingness to sign an informed consent document

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Gaillard, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Women & Infants Center, University of Alabama at Birmingham, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
Started | 8 | 7
Completed | 6 | 6
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Median (Full Range); unit: years] | 43 [35 to 67] | 58 [37 to 83] | 44 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6 | 3 | 9
  Race: Black | 1 | 3 | 4
  Race: Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15
Primary Site Disease [Count of Participants; unit: Participants]
  Cervix, NOS | 4 | 3 | 7
  Endocervix | 4 | 4 | 8
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma (ADC) | 5 | 1 | 6
  Squamous cell (SCC) | 3 | 5 | 8
  Small cell carcinoma + ADC | 0 | 1 | 1
Histology Grade [Count of Participants; unit: Participants]
  Poorly differentiated | 0 | 1 | 1
  Moderately differentiated | 3 | 2 | 5
  Well-differentiated | 2 | 1 | 3
  Unknown/No comment | 3 | 3 | 6
Cervical Cancer Stage [Count of Participants; unit: Participants] — IB -the tumor is 2 centimeters or smaller and the deepest point of tumor invasion is more than 5 millimeters; IIA/IIB-cancer has spread from the cervix to the uterus; IIIC-cancer has spread to the lymph nodes.
  Participants
    IB | 4 | 6 | 10
    IIA/IIB | 3 | 1 | 4
    IIIC | 1 | 0 | 1
Prior Treatment [Count of Participants; unit: Participants]
  Surgery only | 3 | 2 | 5
  ChemoRadiation only | 4 | 3 | 7
  Surgery + ChemoRadiation | 0 | 1 | 1
  Surgery + Radiation | 1 | 1 | 2
Adjuvant Chemo Regimen [Count of Participants; unit: Participants]
  None | 5 | 3 | 8
  Cisplatin | 3 | 3 | 6
  Cisplatin/Etoposide | 0 | 1 | 1
Adjuvant Radiation Site [Count of Participants; unit: Participants]
  No radiation | 3 | 2 | 5
  Cervix | 2 | 1 | 3
  Pelvis involved | 2 | 4 | 6
  Syed brachytherapy | 1 | 0 | 1
Months from end of prior treatment until first vaccination [Median (Full Range); unit: months] | 6.5 [4.5 to 11.6] | 8.4 [4 to 10.9] | 6.7 [4 to 11.6]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility as Assessed by Number of Participants With Treatment-related Adverse Events
Description: Safety and feasibility of intramuscular TA-CIN vaccine via arm or thigh as assessed by number of participants with with a history of HPV16 associated IB1-IV cervical cancer experiencing treatment-emergent adverse events as defined by CTCAE v4.0.
Time Frame: Up to 24 months following the first dose of study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
Number analyzed (Participants) | 8 | 7
Participants
  Treatment-related AEs | 5 | 3
  Treatment-emergent AEs | 8 | 7

2. Secondary Outcome: Antibody Response as Measured by Level of Circulating Antibody in Peripheral Blood
Description: Level of circulating antibody to HPV16 E6, E7, and L2 in the peripheral blood pre- and post-vaccination (visualized by ELISA).
Time Frame: up to 4 years
Population: 1 excluded from efficacy cohort due to withdrawal secondary to toxicity
Measure: Mean (Standard Deviation); unit: absorbance units
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
Number analyzed (Participants) | 7 | 7
absorbance units
  L2-specific antibodies | 1.03 (0.70) | 1.27 (0.92)
  E7-specific antibodies | 0.91 (0.97) | 0.66 (0.78)
  E6-specific antibodies | 0.32 (0.32) | 0.17 (0.17)

3. Secondary Outcome: T-Cell Response as Measured by Level of Circulating T-cells in Peripheral Blood
Description: Level of circulating HPV16 E6- and E7- specific CD8+ T cells and/or CD4+ T cells in the peripheral blood pre- and post-vaccination (visualized by ELISPOT)
Time Frame: up to 4 years
Population: Lack of assay sensitivity for rare T cell populations. Data will not be collected or analyzed in the future.
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mononucleocyte Response
Description: Proliferative responses of peripheral blood mononucleocytes pre- and post-vaccination in response to stimulation by HPV16 E6, E7 and L2
Time Frame: up to 4 years
Population: Blood sample exhaustion. Data will not be collected or analyzed in the future.
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Circulating HPV16 E6-/E7-specific CD8+ T Cells
Description: Levels of circulating HPV16 E6- and E7-specific CD8+ T cells in the peripheral blood pre- and post-vaccination (measured using T-cell receptor sequencing)
Time Frame: up to 4 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Levels of HPV-specific Neutralizing Antibodies
Description: Levels of HPV-specific neutralizing antibodies in the peripheral blood pre- and post-vaccination
Time Frame: up to 4 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Residual HPV16 Viral Load
Description: Residual HPV16 viral load in plasma
Time Frame: 4 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clinical Response as Measured by Time to Disease Recurrence
Description: Clinical response associated with vaccine induced immune responses as measured by Time from administration of TA-CIN to disease recurrence.
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months following the first dose of study vaccine
Description: Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected, recorded, and followed as appropriate.
Arm/Group | TA-CIN Administration Via Thigh | TA-CIN Administration Via Arm
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TA-CIN Administration Via Thigh (N=8) | TA-CIN Administration Via Arm (N=7)
Bowel obstruction (adhesion-related) (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TA-CIN Administration Via Thigh (N=8) | TA-CIN Administration Via Arm (N=7)
Injection site reaction (General disorders) | 5 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General disorders-admin site condition-other (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Investigations (Investigations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Obstruction gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02405221/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02405221/ICF_001.pdf